CLINICAL TRIAL: NCT01914146
Title: Insulin Therapy and Falls Due to Orthostatic Hypotension (Pilot Study)
Brief Title: Insulin Therapy and Falls Due to Orthostatic Hypotension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was changed to Insulin, hypotension and sarcopenia
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kenneth Madden, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H13-01375
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Orthostatic Hypotension; Diabetes; Syncope
Keywords: Diabetes; Insulin; Orthostatic Hypotension; Falls; Syncope
MeSH Terms: conditions — Hypotension, Orthostatic; Diabetes Mellitus; Syncope; Insulin Resistance | interventions — Insulin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before Initiation of Insulin Therapy (Other): Study sessions will occur before the initiation of insulin therapy (no insulin). Initiation of insulin administration will be determined as part of standard of care by the subjects diabetologist in the VGH Diabetes Centre and not as part of participation in this study.
  Interventions: Other: No Insulin
- After Initiation of Insulin Therapy (Other): Study session will take place 2-4 weeks after the initiation of insulin therapy. Initiation of insulin administration will be determined as part of standard of care by the subjects diabetologist in the VGH Diabetes Centre and not as part of participation in this study.
  Interventions: Other: Insulin

INTERVENTIONS:
Other: Insulin — Initiation of insulin administration will be determined as part of standard of care by the subjects diabetologist in the VGH Diabetes Centre and not as part of participation in this study.
  Other Names: Lantus
  Arms: After Initiation of Insulin Therapy
Other: No Insulin — Study session will occur prior to initiation of insulin therapy.
  Arms: Before Initiation of Insulin Therapy

SUMMARY:
In the proposed study, the investigators examine in older adults with Type 2 diabetes the impact of beginning insulin therapy on the orthostatic drop in blood pressure as well as the response of arterial blood pressure and Doppler measures of cerebral blood flow during upright tilt. The investigators hypothesize that in older adults with Type 2 diabetes, the cardiovascular effects of insulin would precipitate or worsen orthostatic intolerance not present at baseline.

DETAILED DESCRIPTION:
Before and 2 weeks after the start of standard insulin therapy several tests will be done:

* orthostatic hypotension will be tested for with 3 orthostatic maneuvers
* vasovagal syncope will be tested with 2 tilt table tests, one augmented with 400ug of nitroglycerin
* MCA velocity will be measured with a transcranial doppler
* Heart Rate and Blood Pressure will be measured throughout the test with a Finometer and Power Lab on a beat to beat basis

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be 65 years of age or older
* All must have been diagnosed with Type 2 diabetes for at least 5 years
* All subjects must be insulin-naïve on recruitment
* All subjects must be eligible to start insulin therapy (long or intermediate acting) as determined by their diabetologist

Exclusion Criteria:

* Anemia, as determined by serum hematocrit
* Abnormal liver function tests
* Elevated creatinine
* Smoker
* Musculoskeletal or neurological condition that would preclude tilt table testing or orthostatic vitals

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
1. Presence or absence of orthostatic hypotension | 1 day
  defined as a drop in systolic blood pressure greater than 20 mmHg after 3 minutes upright standing

SECONDARY OUTCOMES:
1. The nadir of middle cerebral artery (MCA) velocity | 1 day
  lowest middle cerebral artery flow velocity determined by transcranial Doppler
2. The presence or absence of a positive augmented tilt table test | 1 day
  The augmented tilt table test will occur after receiving 300 μg nitroglycerin (GTN), and is a recognized method of testing for risk of vasovagal syncope. The tilt table will be considered positive and aborted prior to the 20 minutes if the subjects have a syncopal spell or demonstrate presyncopal (lightheadedness) symptoms in association with a 30 mm Hg drop in systolic blood pressure.
3. The nadir of systolic blood pressure (SBP) and diastolic blood pressure (DBP) during tilt table test. | 1 day
  lowest systolic blood pressure and diastolic blood pressure during tilt table tests and when they occur.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Madden, MD, Principal Investigator — University of British Columbia
Locations (1):
- Gerontology Research Lab, Dept. of Medicine, Vancouver Coastal Health Research Institute, VGH Research Pavilion, Room 186-828 West 10th Avenue, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No